CLINICAL TRIAL: NCT00967239
Title: The Pharmacogenomics of Breast Cancer Prevention: A Genome-Wide Association Study in Participants Experiencing Breast Cancer Events in High-Risk Postmenopausal Women Receiving Selective Estrogen Receptor Modulators on NSABP Trials P-1 and P-2
Brief Title: Study of Blood Samples From High-Risk Postmenopausal Women Who Received Treatment on Breast Cancer Prevention Clinical Trials NSABP-P-1 or NSABP-P-2
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: NSABP Foundation Inc (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NSABP MCO831; NSABP-MC083I
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Breast Cancer
Keywords: ductal breast carcinoma in situ; invasive ductal breast carcinoma; invasive lobular breast carcinoma; invasive lobular breast carcinoma with predominant in situ component
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Carcinoma, Ductal, Breast; Carcinoma, Lobular | interventions — Amplified Fragment Length Polymorphism Analysis; Pharmacogenomic Testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: None Retained — DNA extracted from stored lymphocytes
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: DNA analysis
Genetic: polymorphism analysis
Other: laboratory biomarker analysis
Other: pharmacogenomic studies

SUMMARY:
RATIONALE: Studying the genes expressed in samples of blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is looking at blood samples from high-risk postmenopausal women who received treatment on breast cancer prevention clinical trials NSABP-P-1 or NSABP-P-2.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To identify genes associated with breast events (i.e., the occurrence of invasive breast cancer or ductal carcinoma in situ), in terms of single-nucleotide polymorphisms (SNPs) in a genome-wide association study, in Caucasian women at high risk of developing breast cancer who have received a selective estrogen receptor modulator (SERM) (i.e., tamoxifen or raloxifene) on the NSABP-P-1 OR NSABP-P-2 breast cancer prevention clinical trials.
* To determine the impact of CYP2D6 metabolizer status, which includes genotype and status of concurrent use of CYP2D6 inhibitors, on breast cancer events in participants receiving either tamoxifen or raloxifene.

Secondary

* To explore whether multiple SNPs within a region are independently associated with a breast event.
* To explore whether there are interactions among SNPs that increase the risk for a breast event.
* To explore whether there is interaction of any SNPs identified in the primary objective with randomized treatment, in terms of the risk for a breast event.
* To identify rare variants that might affect estrogen-dependent expression of chromosomes (CTSO) 4 and 16 (ZNF423) and/or the relationship to BRCA1 expression.

OUTLINE: Samples are stratified according to CYP2D6 genotype and CYP2D6 metabolizer status.

DNA extracted from previously collected blood samples is analyzed in a genome-wide association study and compared with 2 control samples from patients who did not experience a breast event. DNA samples are used to identify and analyze single nucleotide polymorphisms.

Also, exploratory analyses are conducted examining the impact of CYP2D6 metabolizer status on breast cancer events according to invasive vs non-invasive disease, ER status, PgR status, histologic type, and TMN stage.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Previously treated on the NSABP-P-1 Breast Cancer Prevention clinical trial

    * Caucasian women that did or did not experience an invasive breast cancer or ductal carcinoma in situ (DCIS)
    * At least 50 years of age at time of entry to P-1
  * Previously treated on the NSABP-P-2 Breast Cancer Prevention clinical trial

    * Caucasian women that did or did not experience an invasive breast cancer or DCIS
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Postmenopausal status

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: breast cancer cases and matched controls from: participants in NSABP P-1 (tamoxifen or no tamoxifen) participants in NSABP P-2 (raloxifene or no raloxifene; tamoxifen or no tamoxifen)
Sampling Method: Non-Probability Sample
Enrollment: 1881 (Estimated)
Dates: Start 2009-04; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Identification of genes, as measured by single-nucleotide polymorphisms (SNPs), that are associated with breast events | Approximately 6 years
  Retrospective study design: SNPs associated with available breast cancer events
Impact of CYP2D6 metabolizer status on breast cancer events | Approximately 6 years
  Retrospective study design: assay results associated with available breast cancer events

SECONDARY OUTCOMES:
Exploration of whether SNPs within a region are independently associated with a breast event | Approximately 6 years
  Retrospective study design: assay results associated with available breast cancer events
Exploration of whether interactions among SNPs increase the risk for a breast event | Approximately 6 years
  Retrospective study design: results associated with available breast cancer events
Exploration of whether SNPs have an effect on treatment | Approximately 6 years
  Retrospective study design: SNPs associated with appropriate treatment information

CONTACTS AND LOCATIONS:
Overall Officials: James N. Ingle, MD, Study Chair — Mayo Clinic

REFERENCES:
- [Derived] Goetz MP, Schaid DJ, Wickerham DL, Safgren S, Mushiroda T, Kubo M, Batzler A, Costantino JP, Vogel VG, Paik S, Carlson EE, Flockhart DA, Wolmark N, Nakamura Y, Weinshilboum RM, Ingle JN, Ames MM. Evaluation of CYP2D6 and efficacy of tamoxifen and raloxifene in women treated for breast cancer chemoprevention: results from the NSABP P1 and P2 clinical trials. Clin Cancer Res. 2011 Nov 1;17(21):6944-51. doi: 10.1158/1078-0432.CCR-11-0860. Epub 2011 Aug 31. PMID 21880792